CLINICAL TRIAL: NCT04342195
Title: Acquiring Convalescent Specimens to Isolate and Identify Potent Monoclonal Antibodies Against COVID-19
Brief Title: Acquiring Convalescent Specimens for COVID-19 Antibodies
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAS9517
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; Coronavirus Infection; Corona Virus Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood from which peripheral blood mononuclear cells (PBMCs) and plasma will be processed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Blood draw — Participants will have approximately 45 ml of whole blood drawn (3 Tablespoons) drawn at the study visit.

SUMMARY:
Blood samples from participants who have recovered from COVID-19 infection will be obtained and studied. The goal of the research is to identify antibodies that have been generated by the patient to fight the COVID-19 infection. By identifying the most effective antibodies, scientists can make specific antibodies to use to prevent future coronavirus outbreaks or to treat patients with severe disease.

DETAILED DESCRIPTION:
Coronavirus disease (COVID-19), an infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), has caused over 1,273,712 infections and over 69,458 deaths worldwide. Columbia University Irving Medical Center/NewYork-Presbyterian (CUIMC/NYP) has assembled a team of committed virologists, molecular biologists, chemists, and technologists to address this emerging threat. Monoclonal antibodies have become great additions to our therapeutic arsenal, primarily in treating cancer or autoimmune diseases. Recently, the use of monoclonal antibodies in combating infections such as respiratory syncytial virus and HIV have also become clear. In recent years, advanced cell sorting and sequencing technologies have been utilized to identify neutralizing antibodies from human B cells. This protocol will outline our approach to obtaining blood specimens from participants who are recovering from COVID-19 infection. Potential participants will be referred by health care providers from within the CUIMC/NYP system and from outside institutions. If the potential participant agrees to be contacted, study staff will call them to review the informed consent, eligibility criteria and study procedures, and set up a study visit for blood draw. Monoclonal antibodies that could potently neutralize 2019 novel coronavirus (2019-nCoV) and related coronaviruses will be isolated from these specimens. Candidate monoclonal antibodies will then be optimized and evaluated for therapeutic potential. The ultimate goal would be able to produce a monoclonal antibody that could confer protection during an outbreak or be utilized to treat patients with severe COVID disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 (inclusive)
* Confirmed COVID-19 infection by a FDA-approved molecular based assay (including those under emergency use authorization) of respiratory or blood specimens;
* If symptomatic with COVID-19, must have evidence of improvement of symptoms and a duration of at least 4 weeks from the onset of symptoms to day of enrollment;
* If asymptomatic, must have a duration of at least 4 weeks from first positive molecular based COVID-19 assay to day of enrollment

Exclusion Criteria:

* <18 years or >65 years old
* No confirmed diagnosis of COVID-19

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have recovered from COVID-19 infection.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Number of antibodies against coronaviruses isolated and identified from patient samples | Up to 12 months after collection visit
  The blood specimen will be proceeded into peripheral blood mononuclear cells and plasma to be stored for testing. In brief, CD27+ memory B cells that can bind to a SARS-CoV-2 S protein bait will be sorted by flow cytometry and RNA will be extracted to obtain heavy and light chain sequences. Antibody sequences will be annotated using bioinformatics approaches, and candidate sequences will be cloned. Purified antibodies will be characterized and neutralization breadth and potency against SARS-CoV-2 and other related coronaviruses will be assessed using neutralization assays.

CONTACTS AND LOCATIONS:
Overall Officials: David Ho, M.D,, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center/NYP, New York, New York, United States